CLINICAL TRIAL: NCT03517462
Title: Microfilarial Clearance From the Eye and Ocular Changes Associated With Ivermectin Treatment in Individuals With Onchocerciasis
Brief Title: Ocular Changes After Ivermectin - (DOLF IVM/Oncho)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Case Western Reserve University (Other); University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201804116
Record Dates: First submitted 2018-04-23; First posted 2018-05-07 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Onchocerciasis
Keywords: mass drug administration; ophthalmology
MeSH Terms: conditions — Onchocerciasis | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Participants are all given a standard treatment (ivermectin) for onchocerciasis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ivermectin (Experimental): Single dose directly observed treatment with Ivermectin 3Mg Tab (150 ug/kg) delivered orally.
  Interventions: Drug: Ivermectin 3Mg Tab

INTERVENTIONS:
Drug: Ivermectin 3Mg Tab — ivermectin tablet

SUMMARY:
The DOLF Ocular Changes after Ivermectin study will investigate the kinetics of O. volvulus microfilaria (Mf) in the eye following treatment with ivermectin. The primary objective is to determine the proportion of participants with complete Mf clearance from the eye at 3 and 6 months following treatment with ivermectin (IVM).

DETAILED DESCRIPTION:
This study will examine the kinetics of Mf clearance in the eye following ivermectin treatment. Previous studies have been unable to fully assess clearance Mf from the posterior chamber of the eye. This study will be the first to use optical coherence tomography (OCT) in patients with onchocerciasis to document parasites and pathology in the anterior and posterior chambers of the eye, and assess ocular changes following standard ivermectin treatment.

This will be a biomedical prospective cohort study.

The cohort will be stratified based on Mf levels to achieve approximately the following distribution of individuals with roughly one-third of participants in each group.

1. Individuals with positive skin snip Mf density of ≥ 1 Mf/mg), but no observable Mf in eyes using slit lamp and indirect ophthalmoscopy
2. Individuals with positive skin snip Mf density of ≥ 1 Mf/mg and 1-10 Mf in either eye at baseline (based on the highest number counted in either eye)
3. Individuals with positive skin snip Mf density of ≥ 1 Mf/mg and >10 Mf in either eye at baseline.

All participants recruited into the study will be treated with a single dose of ivermectin (150 ug/kg) by mouth under direct observation. This is the standard of care for treatment with onchocerciasis.

Participants will be evaluated following treatment with detailed parasitological and ocular examinations 7 days, 3 months and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 1 palpable subcutaneous nodule (onchocercoma) and ≥ 1 Mf/mg of skin (by skin snip)

Exclusion Criteria:

* Pregnancy and breastfeeding mothers within 1 month of giving birth
* Have base line eye diseases including glaucoma, uveitis, severe keratitis, and/or cataracts that interfere with visualization of the posterior segment of the eye.
* Prior allergic / hypersensitivity reactions or intolerance to ivermectin
* Treatment with ivermectin in the past 6 (six) months

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with complete microfilaria clearance from the eye at 3 months | 3 months following treatment
  Microfilaria in the anterior chamber of the eye will be counted during slit lamp examination at time of assessment. Participants without Mf in the eye will be considered clear of infection in the eye.
Number of participants with complete microfilaria clearance from the eye at 6 months | 6 months following treatment
  Microfilaria in the anterior chamber of the eye will be counted during slit lamp examination at time of assessment. Participants without Mf in the eye will be considered clear of infection in the eye.

SECONDARY OUTCOMES:
The change from baseline in the number of microfilaria detected in the skin at 3 months | baseline, and 3 months following treatment
  Microfilaria (Mf) in the skin will be detected by skin snip microscopy. Up to four (4) skin snips using a corneoscleral punch will be weighed on an analytical balance and incubated for at least 8 hours in isotonic saline in a well of a flat-bottomed microtitre plate at ambient temperature. The Mf that have emerged will be counted using a microscope. Mf number and skin snip weight will be recorded. The mean skin microfilarial density will be calculated and recorded as mf/mg.
The change from baseline in the number of microfilaria detected in the skin at 6 months | baseline, and 6 months following treatment
  Microfilaria (Mf) in the skin will be detected by skin snip microscopy. Up to four (4) skin snips using a corneoscleral punch will be weighed on an analytical balance and incubated for at least 8 hours in isotonic saline in a well of a flat-bottomed microtitre plate at ambient temperature. The Mf that have emerged will be counted using a microscope. Mf number and skin snip weight will be recorded. The mean skin microfilarial density will be calculated and recorded as mf/mg.
The change from baseline in the number of microfilaria detected in the eye at 3 months | baseline, 3 months following treatment
  Microfilaria in the anterior chamber of the eye will be counted during slit lamp examination at time of assessment.
The change from baseline in the number of microfilaria detected in the eye at 6 months | baseline, 6 months following treatment
  Microfilaria in the anterior chamber of the eye will be counted during slit lamp examination at time of assessment.
Number of participants with complete microfilaria clearance from the skin at 3 months | 3 months following treatment
  Microfilaria (Mf) in the skin will be detected by skin snip microscopy. Up to four (4) skin snips using a corneoscleral punch will be weighed on an analytical balance and incubated for at least 8 hours in isotonic saline in a well of a flat-bottomed microtitre plate at ambient temperature. The Mf that have emerged will be counted using a microscope. Mf number and skin snip weight will be recorded. Participants without Mf in the skin will be considered clear of infection in the skin.
Number of participants with complete microfilaria clearance from the skin at 6 months | 6 months following treatment
  Microfilaria (Mf) in the skin will be detected by skin snip microscopy. Up to four (4) skin snips using a corneoscleral punch will be weighed on an analytical balance and incubated for at least 8 hours in isotonic saline in a well of a flat-bottomed microtitre plate at ambient temperature. The Mf that have emerged will be counted using a microscope. Mf number and skin snip weight will be recorded. Participants without Mf in the skin will be considered clear of infection in the skin.

OTHER OUTCOMES:
Assess the utility of optical coherence tomography for evaluating the presence and clearance of Mf in the anterior and posterior segments of the eye. | baseline, 3 and 6 months following treatment
  Results from the optical coherence tomography (OCT) will be compared with slit lamp and other ocular examinations
Evaluate ocular changes between baseline and 3 months following ivermectin treatment using OCT | baseline, and 3 months following treatment
  Results from the optical coherence tomography (OCT) will be compared in participants pre and post treatment
Evaluate ocular changes between baseline and 6 months following ivermectin treatment using OCT | baseline, and 6 months following treatment
  Results from the optical coherence tomography (OCT) will be compared in participants pre and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gary Weil, MD, Principal Investigator — Washington University School of Medicine; Christopher King, MD PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- University of Health and Allied Sciences, Hohoe, Ghana

IPD SHARING:
Plan to Share IPD: Yes
Datasets used for published results will be shared publically through a journal or other open source data repository so that the broader scientific community can access it. Only de-identified data will be shared publicly.

REFERENCES:
- [Background] Herricks JR, Hotez PJ, Wanga V, Coffeng LE, Haagsma JA, Basanez MG, Buckle G, Budke CM, Carabin H, Fevre EM, Furst T, Halasa YA, King CH, Murdoch ME, Ramaiah KD, Shepard DS, Stolk WA, Undurraga EA, Stanaway JD, Naghavi M, Murray CJL. The global burden of disease study 2013: What does it mean for the NTDs? PLoS Negl Trop Dis. 2017 Aug 3;11(8):e0005424. doi: 10.1371/journal.pntd.0005424. eCollection 2017 Aug. No abstract available. PMID 28771480
- [Background] Progress report on the elimination of human onchocerciasis, 2015-2016. Wkly Epidemiol Rec. 2016 Oct 28;91(43):505-14. No abstract available. English, French. PMID 27801998
- [Background] Taylor HR. Onchocerciasis. Int Ophthalmol. 1990 May;14(3):189-94. doi: 10.1007/BF00158317. PMID 2188920
- [Background] Taylor MJ, Awadzi K, Basanez MG, Biritwum N, Boakye D, Boatin B, Bockarie M, Churcher TS, Debrah A, Edwards G, Hoerauf A, Mand S, Matthews G, Osei-Atweneboana M, Prichard RK, Wanji S, Adjei O. Onchocerciasis Control: Vision for the Future from a Ghanian perspective. Parasit Vectors. 2009 Jan 21;2(1):7. doi: 10.1186/1756-3305-2-7. PMID 19154624
- [Background] Komlan K, Vossberg PS, Gantin RG, Solim T, Korbmacher F, Banla M, Padjoudoum K, Karabou P, Kohler C, Soboslay PT. Onchocerca volvulus infection and serological prevalence, ocular onchocerciasis and parasite transmission in northern and central Togo after decades of Simulium damnosum s.l. vector control and mass drug administration of ivermectin. PLoS Negl Trop Dis. 2018 Mar 1;12(3):e0006312. doi: 10.1371/journal.pntd.0006312. eCollection 2018 Mar. PMID 29494606
- [Background] Zimmerman PA, Dadzie KY, De Sole G, Remme J, Alley ES, Unnasch TR. Onchocerca volvulus DNA probe classification correlates with epidemiologic patterns of blindness. J Infect Dis. 1992 May;165(5):964-8. doi: 10.1093/infdis/165.5.964. PMID 1569351
- [Background] Fischer P, Kipp W, Bamuhiga J, Binta-Kahwa J, Kiefer A, Buttner DW. Parasitological and clinical characterization of Simulium neavei-transmitted onchocerciasis in western Uganda. Trop Med Parasitol. 1993 Dec;44(4):311-21. PMID 8134773
- [Background] Dadzie KY, Bird AC, Awadzi K, Schulz-Key H, Gilles HM, Aziz MA. Ocular findings in a double-blind study of ivermectin versus diethylcarbamazine versus placebo in the treatment of onchocerciasis. Br J Ophthalmol. 1987 Feb;71(2):78-85. doi: 10.1136/bjo.71.2.78. PMID 3548811
- [Background] Donnelly JJ, Taylor HR, Young E, Khatami M, Lok JB, Rockey JH. Experimental ocular onchocerciasis in cynomolgus monkeys. Invest Ophthalmol Vis Sci. 1986 Apr;27(4):492-9. PMID 3957567
- [Background] Bird AC, el-Sheikh H, Anderson J, Fuglsang H. Changes in visual function and in the posterior segment of the eye during treatment of onchocerciasis with diethylcarbamazine citrate. Br J Ophthalmol. 1980 Mar;64(3):191-200. doi: 10.1136/bjo.64.3.191. PMID 7387952
- [Background] Duke BO. Human onchocerciasis--an overview of the disease. Acta Leiden. 1990;59(1-2):9-24. PMID 2198761
- [Background] Braun G, McKechnie NM, Connor V, Gilbert CE, Engelbrecht F, Whitworth JA, Taylor DW. Immunological crossreactivity between a cloned antigen of Onchocerca volvulus and a component of the retinal pigment epithelium. J Exp Med. 1991 Jul 1;174(1):169-77. doi: 10.1084/jem.174.1.169. PMID 2056276
- [Background] Chandrashekar R, Curtis KC, Weil GJ. Molecular characterization of a parasite antigen in sera from onchocerciasis patients that is immunologically cross-reactive with human keratin. J Infect Dis. 1995 Jun;171(6):1586-92. doi: 10.1093/infdis/171.6.1586. PMID 7539474
- [Background] Chandrashekar R, Ogunrinade AF, Alvarez RM, Kale OO, Weil GJ. Circulating immune complex-associated parasite antigens in human onchocerciasis. J Infect Dis. 1990 Nov;162(5):1159-64. doi: 10.1093/infdis/162.5.1159. PMID 2230240
- [Background] Greene BM, Gbakima AA, Albiez EJ, Taylor HR. Humoral and cellular immune responses to Onchocerca volvulus infection in humans. Rev Infect Dis. 1985 Nov-Dec;7(6):789-95. doi: 10.1093/clinids/7.6.789. PMID 4070916
- [Background] Johnson TP, Tyagi R, Lee PR, Lee MH, Johnson KR, Kowalak J, Elkahloun A, Medynets M, Hategan A, Kubofcik J, Sejvar J, Ratto J, Bunga S, Makumbi I, Aceng JR, Nutman TB, Dowell SF, Nath A. Nodding syndrome may be an autoimmune reaction to the parasitic worm Onchocerca volvulus. Sci Transl Med. 2017 Feb 15;9(377):eaaf6953. doi: 10.1126/scitranslmed.aaf6953. PMID 28202777
- [Background] Kawabata M, Izui S, Anan S, Kondo S, Fukumoto S, Flores GZ, Kobayakawa T. Circulating immune complexes and their possible relevance to other immunological parameters in Guatemalan onchocerciasis. Int Arch Allergy Appl Immunol. 1983;72(2):128-33. doi: 10.1159/000234854. PMID 6874107
- [Background] Semba RD, Murphy RP, Newland HS, Awadzi K, Greene BM, Taylor HR. Longitudinal study of lesions of the posterior segment in onchocerciasis. Ophthalmology. 1990 Oct;97(10):1334-41. doi: 10.1016/s0161-6420(90)32413-2. PMID 2243684
- [Background] Banla M, Tchalim S, Karabou PK, Gantin RG, Agba AI, Kere-Banla A, Helling-Giese G, Heuschkel C, Schulz-Key H, Soboslay PT. Sustainable control of onchocerciasis: ocular pathology in onchocerciasis patients treated annually with ivermectin for 23 years: a cohort study. PLoS One. 2014 Jun 2;9(6):e98411. doi: 10.1371/journal.pone.0098411. eCollection 2014. PMID 24887413
- [Background] Diawara L, Traore MO, Badji A, Bissan Y, Doumbia K, Goita SF, Konate L, Mounkoro K, Sarr MD, Seck AF, Toe L, Touree S, Remme JH. Feasibility of onchocerciasis elimination with ivermectin treatment in endemic foci in Africa: first evidence from studies in Mali and Senegal. PLoS Negl Trop Dis. 2009 Jul 21;3(7):e497. doi: 10.1371/journal.pntd.0000497. PMID 19621091
- [Background] Traore S, Wilson MD, Sima A, Barro T, Diallo A, Ake A, Coulibaly S, Cheke RA, Meyer RR, Mas J, McCall PJ, Post RJ, Zoure H, Noma M, Yameogo L, Seketeli AV, Amazigo UV. The elimination of the onchocerciasis vector from the island of Bioko as a result of larviciding by the WHO African Programme for Onchocerciasis Control. Acta Trop. 2009 Sep;111(3):211-8. doi: 10.1016/j.actatropica.2009.03.007. Epub 2009 Mar 31. PMID 19619686
- [Background] Rodriguez-Perez MA, Fernandez-Santos NA, Orozco-Algarra ME, Rodriguez-Atanacio JA, Dominguez-Vazquez A, Rodriguez-Morales KB, Real-Najarro O, Prado-Velasco FG, Cupp EW, Richards FO Jr, Hassan HK, Gonzalez-Roldan JF, Kuri-Morales PA, Unnasch TR. Elimination of Onchocerciasis from Mexico. PLoS Negl Trop Dis. 2015 Jul 10;9(7):e0003922. doi: 10.1371/journal.pntd.0003922. eCollection 2015. PMID 26161558
- [Background] Zarroug IM, Hashim K, ElMubark WA, Shumo ZA, Salih KA, ElNojomi NA, Awad HA, Aziz N, Katabarwa M, Hassan HK, Unnasch TR, Mackenzie CD, Richards F, Higazi TB. The First Confirmed Elimination of an Onchocerciasis Focus in Africa: Abu Hamed, Sudan. Am J Trop Med Hyg. 2016 Nov 2;95(5):1037-1040. doi: 10.4269/ajtmh.16-0274. Epub 2016 Jun 27. PMID 27352878
- [Background] Evans DS, Unnasch TR, Richards FO. Onchocerciasis and lymphatic filariasis elimination in Africa: it's about time. Lancet. 2015 May 30;385(9983):2151-2. doi: 10.1016/S0140-6736(15)61022-4. No abstract available. PMID 26068266
- [Background] Fischer PU, King CL, Jacobson JA, Weil GJ. Potential Value of Triple Drug Therapy with Ivermectin, Diethylcarbamazine, and Albendazole (IDA) to Accelerate Elimination of Lymphatic Filariasis and Onchocerciasis in Africa. PLoS Negl Trop Dis. 2017 Jan 5;11(1):e0005163. doi: 10.1371/journal.pntd.0005163. eCollection 2017 Jan. No abstract available. PMID 28056015
- [Background] Kamga GR, Dissak-Delon FN, Nana-Djeunga HC, Biholong BD, Mbigha-Ghogomu S, Souopgui J, Zoure HG, Boussinesq M, Kamgno J, Robert A. Still mesoendemic onchocerciasis in two Cameroonian community-directed treatment with ivermectin projects despite more than 15 years of mass treatment. Parasit Vectors. 2016 Nov 14;9(1):581. doi: 10.1186/s13071-016-1868-8. PMID 27842567
- [Background] Taylor HR, George T. Microfilaria in the cornea in onchocerciasis. Trans R Soc Trop Med Hyg. 1987;81(1):148. doi: 10.1016/0035-9203(87)90308-7. No abstract available. PMID 3445302
- [Background] Wojtkowski M, Bajraszewski T, Gorczynska I, Targowski P, Kowalczyk A, Wasilewski W, Radzewicz C. Ophthalmic imaging by spectral optical coherence tomography. Am J Ophthalmol. 2004 Sep;138(3):412-9. doi: 10.1016/j.ajo.2004.04.049. PMID 15364223
- [Background] Greene BM, Taylor HR, Brown EJ, Humphrey RL, Lawley TJ. Ocular and systemic complications of diethylcarbamazine therapy for onchocerciasis: association with circulating immune complexes. J Infect Dis. 1983 May;147(5):890-7. doi: 10.1093/infdis/147.5.890. PMID 6842023
- [Background] Thomsen EK, Sanuku N, Baea M, Satofan S, Maki E, Lombore B, Schmidt MS, Siba PM, Weil GJ, Kazura JW, Fleckenstein LL, King CL. Efficacy, Safety, and Pharmacokinetics of Coadministered Diethylcarbamazine, Albendazole, and Ivermectin for Treatment of Bancroftian Filariasis. Clin Infect Dis. 2016 Feb 1;62(3):334-341. doi: 10.1093/cid/civ882. Epub 2015 Oct 20. PMID 26486704
- [Background] Greene BM, Taylor HR, Cupp EW, Murphy RP, White AT, Aziz MA, Schulz-Key H, D'Anna SA, Newland HS, Goldschmidt LP, et al. Comparison of ivermectin and diethylcarbamazine in the treatment of onchocerciasis. N Engl J Med. 1985 Jul 18;313(3):133-8. doi: 10.1056/NEJM198507183130301. PMID 3892293
- [Background] Taylor HR, Murphy RP, Newland HS, White AT, D'Anna SA, Keyvan-Larijani E, Aziz MA, Cupp EW, Greene BM. Treatment of onchocerciasis. The ocular effects of ivermectin and diethylcarbamazine. Arch Ophthalmol. 1986 Jun;104(6):863-70. doi: 10.1001/archopht.1986.01050180097039. PMID 3521559
- [Background] Taylor HR, Semba RD, Newland HS, Keyvan-Larijani E, White A, Dukuly Z, Greene BM. Ivermectin treatment of patients with severe ocular onchocerciasis. Am J Trop Med Hyg. 1989 May;40(5):494-500. doi: 10.4269/ajtmh.1989.40.494. PMID 2658637
- [Background] Basanez MG, Pion SD, Boakes E, Filipe JA, Churcher TS, Boussinesq M. Effect of single-dose ivermectin on Onchocerca volvulus: a systematic review and meta-analysis. Lancet Infect Dis. 2008 May;8(5):310-22. doi: 10.1016/S1473-3099(08)70099-9. PMID 18471776
- [Background] Opoku NO, Bakajika DK, Kanza EM, Howard H, Mambandu GL, Nyathirombo A, Nigo MM, Kasonia K, Masembe SL, Mumbere M, Kataliko K, Larbelee JP, Kpawor M, Bolay KM, Bolay F, Asare S, Attah SK, Olipoh G, Vaillant M, Halleux CM, Kuesel AC. Single dose moxidectin versus ivermectin for Onchocerca volvulus infection in Ghana, Liberia, and the Democratic Republic of the Congo: a randomised, controlled, double-blind phase 3 trial. Lancet. 2018 Oct 6;392(10154):1207-1216. doi: 10.1016/S0140-6736(17)32844-1. Epub 2018 Jan 18. PMID 29361335
- [Background] Anderson J, Fuglsang H. Ocular onchocerciasis. Trop Dis Bull. 1977 Apr;74(4):257-72. No abstract available. PMID 329507
- [Background] Anderson J, Fuglsang H. Further studies on the treatment of ocular onchocerciasis with diethylcarbamazine and suramin. Br J Ophthalmol. 1978 Jul;62(7):450-7. doi: 10.1136/bjo.62.7.450. No abstract available. PMID 678497
- [Background] Bird AC, Anderson J, Fuglsang H. Morphology of posterior segment lesions of the eye in patients with onchocerciasis. Br J Ophthalmol. 1976 Jan;60(1):2-20. doi: 10.1136/bjo.60.1.2. PMID 1268156
- [Background] Bird AC, El-Sheikh H, Anderson J, Fuglsang H. Visual loss during oral diethylcarbamazine treatment for onchocerciasis. Lancet. 1979 Jul 7;2(8132):46. doi: 10.1016/s0140-6736(79)90214-9. No abstract available. PMID 87927
- [Background] Fuglsang H, Anderson J. Further observations on the relationship between ocular onchocerciasis and the head nodule, and on the possible benefit of nodulectomy. Br J Ophthalmol. 1978 Jul;62(7):445-9. doi: 10.1136/bjo.62.7.445. PMID 678496
- [Background] Taylor HR. Ivermectin treatment of ocular onchocerciasis. Acta Leiden. 1990;59(1-2):201-6. PMID 2198751
- [Background] Lamberton PH, Cheke RA, Winskill P, Tirados I, Walker M, Osei-Atweneboana MY, Biritwum NK, Tetteh-Kumah A, Boakye DA, Wilson MD, Post RJ, Basanez MG. Onchocerciasis transmission in Ghana: persistence under different control strategies and the role of the simuliid vectors. PLoS Negl Trop Dis. 2015 Apr 21;9(4):e0003688. doi: 10.1371/journal.pntd.0003688. eCollection 2015 Apr. PMID 25897492